CLINICAL TRIAL: NCT01811836
Title: The Effect of Resistant Starch Consumption on Zinc Hemostasis in Malawian Children at Risk for Zinc Deficiency
Brief Title: Zinc Resistant Starch Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201211114
Record Dates: First submitted 2013-03-07; First posted 2013-03-15 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Enteropathy
MeSH Terms: conditions — Intestinal Diseases | interventions — Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Resistant Starch (Experimental): Oral and intravenous zinc stable isotopes. Zinc: 67Zn (>97% enrichment),68Zn (>99% enrichment) and 70Zn (>95% enrichment) Days 1 and 38: children will be administered 40-75 μg of 67Zn through consumed food. At the end of these days, children will be given an intravenous injection of an accurately measured quantity of ~800 μg of 68Zn.
  Days 3-35: resistant starch feeding -- which will be given to mothers and integrated into the food.
  Interventions: Dietary Supplement: Zinc

INTERVENTIONS:
Dietary Supplement: Zinc — Children will have an assessment of zinc homeostasis; each child is given 2 zinc stable isotopes, one by mouth and one intravenously, followed by a stool and urine collection (4 days.) Zinc isotopes are quantified in the feces and urine, values are used to calculate the primary outcome, net zinc balance. An assessment of EE quantitatively measured using the non-invasive site specific sugar absorption test, each child drinks 100 mL of a sugar solution and a urine collection follows. The quantities of non-metabolizable sugars are measured, and the ratio of two of the sugars, lactulose and mannitol, is a measure of environmental enteropathy. Children will receive a dietary supplement, corn starch, modified to reduce its absorption, for 5 weeks, which they will add to their phala. The RS is a standard food and has been used safely in millions of people for years. After taking this RS for 4 weeks both the zinc stable isotope test and the dual sugar absorption test will be repeated.
  Other Names: Zinc Resistant Starch

SUMMARY:
Broad - to examine the result of feeding RS to 3-5 year old rural Malawian children on zinc homeostasis and environmental enteropathy (EE).

Specific -

1. To measure zinc status using a dual zinc stable isotope assay before and after administering resistant starch (RS) in 20 children.
2. To measure intestinal function using a site-specific sugar absorption test before and after administering RS in 20 children.
3. To determine the relationship between RS and zinc homeostasis.
4. To determine the relationship between RS and environmental enteropathy.

DETAILED DESCRIPTION:
A total of 20 (10 M, 10 F) stunted rural Malawian children aged 36-60 months will be studied to determine if there is an effect of feeding RS on zinc homeostasis and environmental enteropathy. These children are at high risk for zinc deficiency and environmental enteropathy by their demographic characteristics. Children will first have a quantitative assessment of zinc homeostasis where each child is given 2 zinc stable isotopes, one by mouth and another intravenously, which is followed by a stool and urine collection of 4 days. Zinc isotopes are quantified in the feces and urine, and these values are used to calculate the primary outcome, net zinc balance. This is followed by an assessment of environmental enteropathy quantitatively measured using the non-invasive site specific sugar absorption test, where each child drinks 100 mL of a sugar solution and a urine collection follows. The quantities of non-metabolizable sugars are measured, and the ratio of two of the sugars, lactulose and mannitol, is a measure of environmental enteropathy. Then the children will receive a dietary supplement, corn starch that has been modified to reduce its dietary absorption, for 5 weeks, which they will add to their phala. The RS is a standard food product that has been used safely in many millions of people for several decades. After taking this RS for 4 weeks both the zinc stable isotope test and the dual sugar absorption test will be repeated on the children to see if they have improved. These results will offer preliminary data as to whether RS might be used effectively on a large scale in the community to alleviate zinc deficiency and/or environmental enteropathy.

ELIGIBILITY:
Inclusion Criteria:

* Any stunted, otherwise healthy child aged 36-60 months living close to the Chipalonga Health Center. Stunting will be defined as height-for-age Z-score (HAZ) < -2. Children will be selected on the basis of having the lowest weight-for-height Z-scores (WHZ), and by dietary surveys on which their caretakers report consuming animal source foods < twice per month. Previous field work indicates about 80% of children are stunted and almost all children consume animal source foods < twice per month.

Exclusion Criteria:

* Children who are not permanent residents in the village. Additionally, children with severe chronic illness such as cerebral palsy, and those who are receiving other supplementary food, or those who are participating in another research study are all ineligible to participate.

Ages: 36 Months to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Net zinc balance | 4 weeks
  Zinc isotopes are quantified in the feces and urine, and these values are used to calculate net zinc balance. taking this RS for 4 weeks both the zinc stable isotope test and the dual sugar absorption test will be repeated on the children to see if they have improved. These results will offer preliminary data as to whether RS might be used effectively on a large scale in the community to alleviate zinc deficiency and/or environmental enteropathy.

SECONDARY OUTCOMES:
Enteropathy Measurement | 4 weeks
  Environmental enteropathy quantitatively measured using the non-invasive site specific sugar absorption test, where each child drinks 100 mL of a sugar solution and a urine collection follows. The quantities of non-metabolizable sugars are measured, and the ratio of two of the sugars, lactulose and mannitol, is a measure of environmental enteropathy.
Weight and Height Changes | 4 weeks (baseline and end)
  Weight and height will be measured initially and at each visit to measure any changes over the period.
  These outcomes will be measured at baseline enrollment and at the end of the study.
Number of participants with adverse events | 4 weeks
  Measure the safety of zinc resistant starch. The RS is a standard food product that has been used safely in many millions of people for several decades.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Manary, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Project Peanut Butter Factory, Blantyre, Malawi

REFERENCES:
- [Background] Manary MJ, Hotz C, Krebs NF, Gibson RS, Westcott JE, Broadhead RL, Hambidge KM. Zinc homeostasis in Malawian children consuming a high-phytate, maize-based diet. Am J Clin Nutr. 2002 Jun;75(6):1057-61. doi: 10.1093/ajcn/75.6.1057. PMID 12036813
- [Background] Manary MJ, Abrams SA, Griffin IJ, Quimper MM, Shulman RJ, Hamzo MG, Chen Z, Maleta K, Manary MJ. Perturbed zinc homeostasis in rural 3-5-y-old Malawian children is associated with abnormalities in intestinal permeability attributed to tropical enteropathy. Pediatr Res. 2010 Jun;67(6):671-5. doi: 10.1203/PDR.0b013e3181da44dc. PMID 20496476
- [Background] Sazawal S, Bentley M, Black RE, Dhingra P, George S, Bhan MK. Effect of zinc supplementation on observed activity in low socioeconomic Indian preschool children. Pediatrics. 1996 Dec;98(6 Pt 1):1132-7. PMID 8951265
- [Background] Menzies IS, Zuckerman MJ, Nukajam WS, Somasundaram SG, Murphy B, Jenkins AP, Crane RS, Gregory GG. Geography of intestinal permeability and absorption. Gut. 1999 Apr;44(4):483-9. doi: 10.1136/gut.44.4.483. PMID 10075954
- [Background] Sazawal S, Black RE, Bhan MK, Bhandari N, Sinha A, Jalla S. Zinc supplementation in young children with acute diarrhea in India. N Engl J Med. 1995 Sep 28;333(13):839-44. doi: 10.1056/NEJM199509283331304. PMID 7651474
- [Background] Ruel MT, Rivera JA, Santizo MC, Lonnerdal B, Brown KH. Impact of zinc supplementation on morbidity from diarrhea and respiratory infections among rural Guatemalan children. Pediatrics. 1997 Jun;99(6):808-13. doi: 10.1542/peds.99.6.808. PMID 9164774
- [Background] Yonekura L, Suzuki H. Effects of dietary zinc levels, phytic acid and resistant starch on zinc bioavailability in rats. Eur J Nutr. 2005 Sep;44(6):384-91. doi: 10.1007/s00394-004-0540-9. Epub 2004 Nov 23. PMID 16151969
- [Background] Turnlund JR. The use of stable isotopes in mineral nutrition research. J Nutr. 1989 Jan;119(1):7-14. doi: 10.1093/jn/119.1.7. PMID 2643698
- [Background] Miller LV, Hambidge KM, Naake VL, Hong Z, Westcott JL, Fennessey PV. Size of the zinc pools that exchange rapidly with plasma zinc in humans: alternative techniques for measuring and relation to dietary zinc intake. J Nutr. 1994 Feb;124(2):268-76. doi: 10.1093/jn/124.2.268. PMID 8308576
- [Background] Meddings JB, Gibbons I. Discrimination of site-specific alterations in gastrointestinal permeability in the rat. Gastroenterology. 1998 Jan;114(1):83-92. doi: 10.1016/s0016-5085(98)70636-5. PMID 9428222
- [Background] Galpin L, Manary MJ, Fleming K, Ou CN, Ashorn P, Shulman RJ. Effect of Lactobacillus GG on intestinal integrity in Malawian children at risk of tropical enteropathy. Am J Clin Nutr. 2005 Nov;82(5):1040-5. doi: 10.1093/ajcn/82.5.1040. PMID 16280436
- [Result] May T, Westcott C, Thakwalakwa C, Ordiz MI, Maleta K, Westcott J, Ryan K, Hambidge KM, Miller LV, Young G, Mortimer E, Manary MJ, Krebs NF. Resistant starch does not affect zinc homeostasis in rural Malawian children. J Trace Elem Med Biol. 2015 Apr;30:43-48. doi: 10.1016/j.jtemb.2015.01.005. Epub 2015 Jan 21. PMID 25744509
- [Derived] Ordiz MI, May TD, Mihindukulasuriya K, Martin J, Crowley J, Tarr PI, Ryan K, Mortimer E, Gopalsamy G, Maleta K, Mitreva M, Young G, Manary MJ. The effect of dietary resistant starch type 2 on the microbiota and markers of gut inflammation in rural Malawi children. Microbiome. 2015 Sep 3;3:37. doi: 10.1186/s40168-015-0102-9. PMID 26334878